CLINICAL TRIAL: NCT04308499
Title: Pilot Randomized Controlled Trial of Digital Cognitive-Behavioral Therapy for Insomnia in HIV-Infected Individuals
Brief Title: Digital Behavioral Therapy for Sleep Problems
Acronym: dBTS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty to recruit HIV patients with insomnia
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Joshua Hyong-Jin Cho, Associate professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-000064
Record Dates: First submitted 2020-03-09; First posted 2020-03-16 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital cognitive-behavioral therapy for insomnia (dCBTI) (Experimental): Internet-based cognitive-behavioral therapy for insomnia (CBT-I) structured into 6 weekly sessions
  Interventions: Behavioral: Digital cognitive-behavioral therapy for insomnia (dCBTI)
- Sleep hygiene education (SHE) (Active Comparator): Recognized and commonly prescribed set of sleep hygiene instructions
  Interventions: Behavioral: Sleep hygiene education (SHE)

INTERVENTIONS:
Behavioral: Digital cognitive-behavioral therapy for insomnia (dCBTI) — Internet-based cognitive-behavioral therapy for insomnia (CBT-I) structured into 6 weekly sessions accessed using either a computer or a smartphone
  Arms: Digital cognitive-behavioral therapy for insomnia (dCBTI)
Behavioral: Sleep hygiene education (SHE) — Recognized and commonly prescribed set of sleep hygiene instructions comprised of comprise a website and a downloadable booklet
  Arms: Sleep hygiene education (SHE)

SUMMARY:
Insomnia is very common, especially in HIV population (up to 73%), and contributes to the development of other conditions such as depression, dementia, inflammation, obesity, and heart diseases. Cognitive-behavioral therapy for insomnia (CBT-I) is known to improve insomnia. However, it has never been tested in HIV-positive patients. The investigators aim to examine the Internet version of this therapy in HIV-positive patients because the availability of CBT-I is very limited while the cost is high. The investigators will test this internet version, also called digital CBT-I (dCBTI), against sleep hygiene education (SHE), a commonly prescribed set of instructions in clinical practice, in 60 HIV-positive patients with insomnia invited from the Multicenter AIDS Cohort Study (MACS) Los Angeles site. The investigators aim to test if dCBTI or SHE improves insomnia in this patient group. This trial involves a behavioral treatment that can be done from home with minimal side effects and includes neither medications nor invasive interventions. Lastly, this trial will provide important pilot data for a larger trial testing long-term effects of insomnia treatment in HIV-positive patients.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of insomnia disorder
* Aged 18 years or older
* Reliable Internet access using either computer or smartphone
* Ability to read and understand English

Exclusion Criteria:

* High risk of obstructive sleep apnea
* Diagnosis of restless legs syndrome
* Severe health issues requiring hospital admission
* Currently receiving psychological treatment for insomnia
* Reporting current suicidal ideation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) | Weeks 0, 4, 8, and 24
  Change in insomnia severity assessed by a scale with higher scores indicating worse outcome (range 0-28)
Change in Sleep Efficiency | Weeks 0, 4, 8, and 24
  Change in sleep efficiency estimated using sleep diary with higher percentages indicating better outcome (range 0-100%)

SECONDARY OUTCOMES:
Change in Total Sleep Time (TST) | Weeks 0, 4, 8, and 24
  Change in sleep duration
Change in Epworth Sleepiness Scale (ESS) | Weeks 0, 4, 8, and 24
  Change in daytime sleepiness assessed by a scale with higher scores indicating worse outcome (range 0-24)
Change in Center for Epidemiologic Studies Depression Scale (CES-D) | Weeks 0, 4, 8, and 24
  Change in depressive symptoms assessed by a scale with higher scores indicating worse outcome (range 0-60)
Change in Generalized Anxiety Disorder 7-item scale (GAD-7) | Weeks 0, 4, 8, and 24
  Change in anxiety symptoms assessed by a scale with higher scores indicating worse outcome (range 0-21)
Change in Snaith-Hamilton Pleasure Scale (SHAPS) | Weeks 0, 4, 8, and 24
  Change in anhedonia assessed by a scale with higher scores indicating worse outcome (range 0-14)
Change in Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF) | Weeks 0, 4, 8, and 24
  Change in fatigue assessed by a scale with higher scores indicating worse outcome (range 0-120)
Change in UCLA Loneliness Scale (ULS) | Weeks 0, 4, 8, and 24
  Change in loneliness assessed by a scale with higher scores indicating worse outcome (range 20-80)
Change in Insomnia Caseness | Weeks 0, 4, 8, and 24
  Change in probable diagnosis of insomnia assessed using Sleep Condition Indicator (SCI)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Cousins Center for Psychoneuroimmunology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No